CLINICAL TRIAL: NCT06016556
Title: A Retrospective Observational Non-Interventional Study (NIS) to Assess Patient Characteristics and Healthcare Resource Use (HCRU) Among COVID-19 Patients Receiving Treatment With Nirmatrelvir; Ritonavir (PAXLOVID TM) in the Kingdom of Saudi Arabia (KSA).
Brief Title: A Study of COVID-19 Patients Receiving Treatment With Nirmatrelvir; Ritonavir in the Kingdom of Saudi Arabia
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C4671054; NCT06016556 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2023-08-25; First posted 2023-08-29 (Actual); Results first posted 2025-04-29 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Covid-19
Keywords: Paxlovid; Saudi Arabia
MeSH Terms: conditions — COVID-19 | interventions — nirmatrelvir and ritonavir drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Patients receiving Nirmatrelvir; Ritonavir (PAXLOVID): Adult COVID-19 patients' HCRU within the 30-day period following nirmatrelvir, ritonavir prescription.
  Interventions: Drug: nirmatrelvir, ritonavir

INTERVENTIONS:
Drug: nirmatrelvir, ritonavir — single cohort
  Other Names: Paxlovid

SUMMARY:
The aim of this study is to describe the baseline demographic, clinical characteristics, and Healthcare Resource Use (HCRU) of adult (≥18 years) COVID-19 patients who have been prescribed nirmatrelvir, ritonavir treatment.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed COVID-19 infection during the study observation period
* Nirmatrelvir, ritonavir written prescription

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will involve collection of pre-defined, structured data retrospectively from medical records (electronic and/or paper if necessary) of patients who meet the study eligibility criteria and who have been prescribed nirmatrelvir, ritonavir treatment within a 15-month lookback period from the date of site initiation (Cohort 1). The lookback period will span from 01 April 2022 to 30 June 2023. Data abstracted from patients' medical records will include patient demographics and clinical characteristics at index date (defined as the date of nirmatrelvir, ritonavir treatment prescribing), in addition to patients' HCRU during the 30-day period post-index date.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2023-10-17 (Actual); Primary Completion 2024-04-09 (Actual); Study Completion 2024-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- Saudi Arabia (3):
  - King Faisal Specialist Hospital & research center - Jeddah, Jeddah
  - King Abdulaziz Medical City, Riyadh
  - King Faisal Specialist Hospital and Research Center, Riyadh

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4671054

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants who were prescribed nirmatrelvir, ritonavir (PAXLOVIDTM) in the Kingdom of Saudi Arabia (KSA) any day between 1-Apr-2022 to 30-Jun-2023 (15-month look back period) for corona virus disease 2019 (COVID-19) caused by severe acute respiratory syndrome coronavirus (SARSCoV-2)- their data was included in this retrospective observational study.
Pre-assignment Details: Data was extracted from medical records of the participants and data was evaluated per objectives of this study in approximately 6 months of this study (study start date: 17-Oct-2023 to study completion date: 09-Apr-2024).
Groups:
- All Participants: Eligible participants who had COVID-19 and were prescribed nirmatrelvir, ritonavir treatment (PAXLOVIDTM) in KSA- their data was studied retrospectively as per objectives of this study. No intervention was administered to the participants under this study.
Period: Overall Study
Arm/Group | All Participants
Started | 248
Completed | 248
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all eligible participants whose data were included and observed in this study.
Arm/Group | All Participants
Number analyzed (Participants) | 248
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.85 (18.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148
  Male | 100
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Arab | 247
  Ethnicity: Asian/Pacific Islander | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Classified According to Education Level at Index Date
Description: Education level classification: no formal education, primary school, secondary school, undergraduate university degree, master's degree and Doctor of Philosophy (PhD) or doctorate. Index date was defined as the date of nirmatrelvir, ritonavir (PAXLOVIDTM) treatment prescription, which could be any day between 1-Apr-2022 to 30-Jun-2023 (15-month look back period).
Time Frame: At index date; retrospective data was evaluated during approximately 6 months of this study
Population: Analysis population included all eligible participants whose data were included and observed in this study. Here, "Overall Number of Participants Analyzed" signifies those number of participants who had non-missing values and were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 140
Participants
  No formal education | 32
  Primary school | 1
  Secondary school | 22
  Undergraduate university degree | 85
  Master's degree | 0
  PhD or doctorate | 0

2. Primary Outcome: Number of Participants Classified According to Employment Status at Index Date
Description: Employment status classification: full-time employment, part-time employment, homemaker, retired, student, disabled/too ill to work, and unemployed. Index date was defined as the date of nirmatrelvir, ritonavir (PAXLOVIDTM) treatment prescription, which could be any day between 1-Apr-2022 to 30-Jun-2023 (15-month look back period).
Time Frame: At index date; retrospective data was evaluated during approximately 6 months of this study
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 150
Participants
  Full-time employment | 41
  Part-time employment | 1
  Homemaker | 10
  Retired | 42
  Student | 11
  Disabled/too ill to work | 3
  Unemployed | 42

3. Primary Outcome: Height at Index Date
Description: Index date was defined as the date of nirmatrelvir, ritonavir (PAXLOVIDTM) treatment prescription, which could be any day between 1-Apr-2022 to 30-Jun-2023 (15-month look back period).
Time Frame: At index date; retrospective data was evaluated during approximately 6 months of this study
Population: Analysis population included all eligible participants whose data were included and observed in this study. Here, ''Overall Number of Participants Analyzed'' signifies number of participants who had non-missing values and were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | All Participants
Number analyzed (Participants) | 240
Meters | 1.62 (0.10)

4. Primary Outcome: Weight at Index Date
Description: as for outcome 3
Time Frame: At index date; retrospective data was evaluated during approximately 6 months of this study
Population: Analysis population included all eligible participants whose data were included and observed in this study. Here, ''Overall Number of Participants Analyzed'' signifies number of participants who had non-missing values and evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | All Participants
Number analyzed (Participants) | 242
Kilograms | 74.13 (18.81)

5. Primary Outcome: Body Mass Index (BMI) at Index Date
Description: BMI was calculated based on the reported weight and height in the unit of kilograms over squared meters (kg/m^2). Index date was defined as the date of nirmatrelvir, ritonavir (PAXLOVIDTM) treatment prescription, which could be any day between 1-Apr-2022 to 30-Jun-2023 (15-month look back period).
Time Frame: At index date; retrospective data was evaluated during approximately 6 months of this study
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Kg/m^2
Arm/Group | All Participants
Number analyzed (Participants) | 237
Kg/m^2 | 28.25 (6.74)

6. Primary Outcome: Number of Participants Classified According to Smoking Status at Index Date
Description: Smoking status classification: current smoker, former smoker and never smoker. Index date was defined as the date of nirmatrelvir, ritonavir (PAXLOVIDTM) treatment prescription, which could be any day between 1-Apr-2022 to 30-Jun-2023 (15-month look back period).
Time Frame: At index date; retrospective data was evaluated during approximately 6 months of this study
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 222
Participants
  Current smoker | 8 [lower limit 0.10]
  Former smoker | 7 [lower limit 0.10]
  Never smoker | 207 [lower limit 0.10]

7. Primary Outcome: Number of Participants Who Had at Least 1 Pre-existing Comorbidity at Index Date
Description: as for outcome 3
Time Frame: At index date; retrospective data was evaluated during approximately 6 months of this study
Population: Analysis population included all eligible participants whose data were included and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 248
Participants | 224

8. Primary Outcome: Number of Participants Who Had at Least 1 Concomitant Medication for Comorbidities at Index Date
Description: as for outcome 3
Time Frame: At index date; retrospective data was evaluated during approximately 6 months of this study
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 223
Participants | 186

9. Primary Outcome: Number of Participants With COVID-19 Infection During the Last 6 Months Prior to Index Date
Description: as for outcome 3
Time Frame: During 6 months prior to index date, information obtained at index date; retrospective data was evaluated during approximately 6 months of this study
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 246
Participants | 9

10. Primary Outcome: Duration Between Last COVID-19 Infection and Index Date
Description: Duration (in months) between COVID-19 infection in last 6 months prior to index date and index date was reported in this outcome measure. Index date was defined as the date of nirmatrelvir, ritonavir (PAXLOVIDTM) treatment prescription, which could be any day between 1-Apr-2022 to 30-Jun-2023 (15-month look back period).
Time Frame: From 6 months prior to index date up to index date, information obtained at index date; retrospective data was evaluated during approximately 6 months of this study
Population: Analysis population included all eligible participants whose data were included and observed in this study. Here, ''Overall Number of Participants Analyzed'' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | All Participants
Number analyzed (Participants) | 9
Months | 3.34 (2.06)

11. Primary Outcome: Number of Participants Who Had Previously Received at Least 1 Dose of Any COVID-19 Vaccine
Description: as for outcome 3
Time Frame: Historic information obtained at index date; retrospective data was evaluated during approximately 6 months of this study
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 233
Participants | 200 [lower limit 2.06]

12. Primary Outcome: Number of Participants Classified According to the Type of COVID-19 Vaccine Received Previously
Description: One participant could have received more than one type of vaccine. Index date was defined as the date of nirmatrelvir, ritonavir (PAXLOVIDTM) treatment prescription, which could be any day between 1-Apr-2022 to 30-Jun-2023 (15-month look back period).
Time Frame: as for outcome 11
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 147
Participants
  Protein-Serum Institute of India | 1 [lower limit 2.06]
  RNA-Moderna | 1
  RNA-Pfizer/BioNTech | 143
  Viral Vector-Oxford/AstraZeneca | 19

13. Primary Outcome: Duration Between Previous COVID-19 Vaccination Date and Index Date
Description: Duration (in months) between vaccination date and index date was calculated as (index date - date of first covid-19 vaccination date)/30.42. Index date was defined as the date of nirmatrelvir, ritonavir (PAXLOVIDTM) treatment prescription, which could be any day between 1-Apr-2022 to 30-Jun-2023 (15-month look back period).
Time Frame: From date of first COVID-19 vaccination to index date, information obtained at index date; retrospective data was evaluated during approximately 6 months of this study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | All Participants
Number analyzed (Participants) | 142
Months | 23.16 (8.59)

14. Primary Outcome: Number of Participants Classified According to Total Number of Previous COVID-19 Vaccine Doses Taken
Description: as for outcome 3
Time Frame: as for outcome 11
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 146
Participants
  1 | 10
  2 | 45
  3 | 84
  4 | 7

15. Primary Outcome: Number of Participants Classified According to Dose of Nirmatrelvir/Ritonavir Received at Index Date
Description: Classification: 1) Nirmatrelvir at a dose of 300 milligrams (mg), as 2 split doses of 150 mg and Ritonavir at a dose of 100 mg; 2) Other: Nirmatrelvir at a dose of 150 mg, and Ritonavir at a dose of 100 mg. Index date was defined as the date of nirmatrelvir, ritonavir (PAXLOVIDTM) treatment prescription, which could be any day between 1-Apr-2022 to 30-Jun-2023 (15-month look back period).
Time Frame: At index date; retrospective data was evaluated during approximately 6 months of this study
Population: Analysis population included all eligible participants whose data were included and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 248
Participants
  300 mg (2*150)/100 mg | 229
  Other (150 mg/100 mg) | 19

16. Primary Outcome: Number of Participants Classified According to Frequency of Dosing of Nirmatrelvir/Ritonavir (PAXLOVIDTM) at Index Date
Description: Classification: 1) Nirmatrelvir at a dose of 300 mg, as 2 split doses of 150 mg and Ritonavir at a dose of 100 mg; 2) Other: Nirmatrelvir at a dose of 150 mg, and Ritonavir at a dose of 100 mg. Index date was defined as the date of nirmatrelvir, ritonavir (PAXLOVIDTM) treatment prescription, which could be any day between 1-Apr-2022 to 30-Jun-2023 (15-month look back period).
Time Frame: At index date; retrospective data was evaluated during approximately 6 months of this study
Population: Analysis population included all eligible participants whose data were included and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 248
Participants
  Twice a day | 245
  Once | 2
  Once a day on Day 1, then 150mg/100mg once daily on Days 2-5 | 1

17. Primary Outcome: Number of Participants Classified According to Dispensed Type of Nirmatrelvir/Ritonavir (PAXLOVIDTM) at Index Date
Description: Classification of dispensed type: blister, box, tablets. Index date was defined as the date of nirmatrelvir, ritonavir (PAXLOVIDTM) treatment prescription, which could be any day between 1-Apr-2022 to 30-Jun-2023 (15-month look back period).
Time Frame: At index date; retrospective data was evaluated during approximately 6 months of this study
Population: Analysis population included all eligible participants whose data were included and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 248
Participants
  Box | 236
  Tablets | 11
  Blister | 1

18. Primary Outcome: Number of Participants Classified According to Medications Used to Treat COVID-19 Infection at Index Date
Description: Number of participants classified according to medications (apart from Nirmatrelvir/Ritonavir [PAXLOVIDTM]) used to treat COVID-19 infection at index date were reported in this outcome measure. A participant may receive more than one medication to treat COVID-19 infection. Index date was defined as the date of nirmatrelvir, ritonavir (PAXLOVIDTM) treatment prescription, which could be any day between 1-Apr-2022 to 30-Jun-2023 (15-month look back period).
Time Frame: At index date; retrospective data was evaluated during approximately 6 months of this study
Population: Analysis population included all eligible participants whose data were included and observed in this study. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 94
Participants
  Antibiotic: Ceftriaxone | 13
  Antibiotic: Azithromycin | 11
  Antibiotic: Cefepime | 8
  Antibiotic: Vancomycin | 7
  Antibiotic: Meropenem | 5
  Antibiotic: Ceftazidime | 3
  Antibiotic: Amoxicillin | 2
  Antibiotic: Ciprofloxacin | 1
  Antibiotic: Doxycycline | 1
  Antibiotic: Levofloxacin | 1
  Antibiotic: Piperacillin/Tazobactam | 11
  Antiviral: Remdesivir | 39
  Antiviral: Acyclovir | 2
  Antiviral: Oseltamivir | 1
  Steroid: Dexamethasone | 16
  Steroid: Hydrocortisone | 1
  Steroid: Methylprednisolone Sodium Succinate | 1
  Steroid: Prednisolone/ Prednisone | 1
  Steroid: Seretide | 1
  Monoclonal antibody: Tocilizumab | 1
  Antipyretics: Acetaminophen | 3
  Antifungals: Noxafil | 1
  Antifungals: Fluconazole | 1
  Other medications: Esomeprazole | 2
  Other medications: Azathioprine | 2
  Other medications: Cyclosporin | 1
  Other medications: Omeprazole | 1

19. Primary Outcome: Number of Participants Who Were Hospitalized at Index Date
Description: In this outcome measure those number of participants are reported who were prescribed Nirmatrelvir/Ritonavir (PAXLOVIDTM) while they were hospitalized (related or non-related to COVID-19). Index date was defined as the date of nirmatrelvir, ritonavir (PAXLOVIDTM) treatment prescription, which could be any day between 1-Apr-2022 to 30-Jun-2023 (15-month look back period).
Time Frame: Information obtained at index date; retrospective data was evaluated during approximately 6 months of this study
Population: Analysis population included all eligible participants whose data were included and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 248
Participants | 120

20. Primary Outcome: Number of Participants Who Were Hospitalized Due to COVID-19 at Index Date
Description: In this outcome measure those number of participants are reported who were prescribed Nirmatrelvir/Ritonavir (PAXLOVIDTM) while they were hospitalized (related to COVID-19). Index date was defined as the date of nirmatrelvir, ritonavir (PAXLOVIDTM) treatment prescription, which could be any day between 1-Apr-2022 to 30-Jun-2023 (15-month look back period).
Time Frame: Information obtained at index date; retrospective data was evaluated during approximately 6 months of this study
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 120
Participants | 72

21. Primary Outcome: Length of Hospitalization Stay Due to COVID-19 at Index Date
Description: Length of hospitalization stay was measured in days from day of hospitalization (related to COVID-19) till index date. Index date was defined as the date of nirmatrelvir, ritonavir (PAXLOVIDTM) treatment prescription, which could be any day between 1-Apr-2022 to 30-Jun-2023 (15-month look back period).
Time Frame: From day of hospitalization till index date, information obtained at index date; retrospective data was evaluated during approximately 6 months of this study
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | All Participants
Number analyzed (Participants) | 72
Days | 6.64 (6.69)

22. Primary Outcome: Number of Participants With Intensive Care Unit (ICU) Admission at Index Date
Description: In this outcome measure those number of participants are reported who were admitted to ICU while they were prescribed Nirmatrelvir/Ritonavir (PAXLOVIDTM). Index date was defined as the date of nirmatrelvir, ritonavir (PAXLOVIDTM) treatment prescription, which could be any day between 1-Apr-2022 to 30-Jun-2023 (15-month look back period).
Time Frame: Information obtained at index date; retrospective data was evaluated during approximately 6 months of this study
Population: Analysis population included all eligible participants whose data were included and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 248
Participants | 17 [lower limit 6.69]

23. Primary Outcome: Length of ICU Stay Due to COVID-19 at Index Date
Description: Length of ICU stay was measured in days from day of ICU admission till index date. Index date was defined as the date of nirmatrelvir, ritonavir (PAXLOVIDTM) treatment prescription, which could be any day between 1-Apr-2022 to 30-Jun-2023 (15-month look back period).
Time Frame: From day of ICU admission till index date, information obtained at index date; retrospective data was evaluated during approximately 6 months of this study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | All Participants
Number analyzed (Participants) | 6
Days | 17.83 (11.41)

24. Primary Outcome: Number of Participants Who Were on Supplemental Oxygen Use at Index Date
Description: In this outcome measure those number of participants are reported who were on supplemental oxygen use when they were prescribed Nirmatrelvir/Ritonavir (PAXLOVIDTM). Index date was defined as the date of nirmatrelvir, ritonavir (PAXLOVIDTM) treatment prescription, which could be any day between 1-Apr-2022 to 30-Jun-2023 (15-month look back period).
Time Frame: At index date; retrospective data was evaluated during approximately 6 months of this study
Population: Analysis population included all eligible participants whose data were included and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 248
Participants | 14 [lower limit 6.69]

25. Primary Outcome: Number of Participants Who Were on Vasopressor Use at Index Date
Description: In this outcome measure those number of participants are reported who were on vasopressor use when they were prescribed Nirmatrelvir/Ritonavir (PAXLOVIDTM). Index date was defined as the date of nirmatrelvir, ritonavir (PAXLOVIDTM) treatment prescription, which could be any day between 1-Apr-2022 to 30-Jun-2023 (15-month look back period).
Time Frame: At index date; retrospective data was evaluated during approximately 6 months of this study
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 120
Participants | 0 [lower limit 6.69]

26. Primary Outcome: Number of Participants With Intubation at Index Date
Description: In this outcome measure those number of participants are reported who were intubated when they were prescribed Nirmatrelvir/Ritonavir (PAXLOVIDTM). Index date was defined as the date of nirmatrelvir, ritonavir (PAXLOVIDTM) treatment prescription, which could be any day between 1-Apr-2022 to 30-Jun-2023 (15-month look back period).
Time Frame: At index date; retrospective data was evaluated during approximately 6 months of this study
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 120
Participants | 2 [lower limit 6.69]

27. Primary Outcome: Number of Participants With Outpatient Visits at Index Date
Description: as for outcome 3
Time Frame: At index date; retrospective data was evaluated during approximately 6 months of this study
Population: Analysis population included all eligible participants whose data were included and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 248
Participants | 32 [lower limit 6.69]

28. Primary Outcome: Number of Participants Who Had Emergency Room (ER) Visits Due to COVID-19 at Index Date
Description: as for outcome 3
Time Frame: At index date; retrospective data was evaluated during approximately 6 months of this study
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 146
Participants | 126 [lower limit 6.69]

29. Secondary Outcome: Number of Participants Who Were Hospitalized During the 30-day Post-Index Period
Description: as for outcome 3
Time Frame: 30-day post index date; retrospective data was evaluated during approximately 6 months of this study
Population: Analysis population included all eligible participants whose data were included and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 248
Participants | 23 [lower limit 6.69]

30. Secondary Outcome: Number of Participants Who Were Hospitalized Due to COVID-19 During the 30-day Post-Index Period
Description: as for outcome 3
Time Frame: 30-day post index date; retrospective data was evaluated during approximately 6 months of this study
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 23
Participants | 2 [lower limit 6.69]

31. Secondary Outcome: Length of Hospitalization Stay Due to COVID-19 During the 30-day Post-Index Period
Description: as for outcome 3
Time Frame: 30-day post index date; retrospective data was evaluated during approximately 6 months of this study
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | All Participants
Number analyzed (Participants) | 2
Days | 23.00 (26.87)

32. Secondary Outcome: Number of Participants With ICU Admission During the 30-day Post-Index Period
Description: as for outcome 3
Time Frame: 30-day post index date; retrospective data was evaluated during approximately 6 months of this study
Population: Analysis population included all eligible participants whose data were included and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 248
Participants | 9 [lower limit 26.87]

33. Secondary Outcome: Length of ICU Stay Due to COVID-19 During the 30-day Post-Index Period
Description: as for outcome 3
Time Frame: 30-day post index date; retrospective data was evaluated during approximately 6 months of this study
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | All Participants
Number analyzed (Participants) | 2
Days | 8.00 (7.07)

34. Secondary Outcome: Number of Participants Who Were on Supplemental Oxygen Use During the 30-day Post-Index Period
Description: as for outcome 3
Time Frame: 30-day post index date; retrospective data was evaluated during approximately 6 months of this study
Population: Analysis population included all eligible participants whose data were included and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 248
Participants | 6 [lower limit 7.07]

35. Secondary Outcome: Number of Participants Who Were on Vasopressor Use During the 30-day Post-Index Period
Description: as for outcome 3
Time Frame: 30-day post index date; retrospective data was evaluated during approximately 6 months of this study
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 23
Participants | 1 [lower limit 7.07]

36. Secondary Outcome: Number of Participants With Intubation During the 30-day Post-Index Period
Description: as for outcome 3
Time Frame: 30-day post index date; retrospective data was evaluated during approximately 6 months of this study
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 23
Participants | 2 [lower limit 7.07]

37. Secondary Outcome: Number of Participants Who Had Outpatient Visits During the 30-day Post-Index Period
Description: as for outcome 3
Time Frame: 30-day post index date; retrospective data was evaluated during approximately 6 months of this study
Population: Analysis population included all eligible participants whose data were included and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 248
Participants | 61 [lower limit 7.07]

38. Secondary Outcome: Number of Participants Who Had ER Visits Due to COVID-19 During the 30-day Post-Index Period
Description: as for outcome 3
Time Frame: 30-day post index date; retrospective data was evaluated during approximately 6 months of this study
Population: Analysis population included all eligible participants whose data were included and observed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 248
Participants | 21 [lower limit 7.07]

39. Secondary Outcome: Number of Participants Classified According to COVID-19 Polymerase Chain Reaction (PCR) and Antigen Test Results During the 30-day Post-Index Period
Description: as for outcome 3
Time Frame: 30-day post index date; retrospective data was evaluated during approximately 6 months of this study
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 17
Participants
  Antigen-Negative | 4 [lower limit 7.07]
  Antigen-Positive | 1 [lower limit 7.07]
  PCR-Negative | 7 [lower limit 7.07]
  PCR-Positive | 5 [lower limit 7.07]

40. Secondary Outcome: Time to Negative COVID-19 Test During the 30-day Post-Index Period
Description: Index date was defined as the date of nirmatrelvir, ritonavir (PAXLOVIDTM) treatment prescription, which could be any day between 1-Apr-2022 to 30-Jun-2023 (15-month look back period). Time to negative COVID-19 test was assessed from index date till participant tested negative for COVID-19 during 30 days post index period.
Time Frame: 30-day post index date; retrospective data was evaluated during approximately 6 months of this study
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | All Participants
Number analyzed (Participants) | 11
Days | 15.09 (11.13)

ADVERSE EVENTS:
Time Frame: From Index date up to 30 days post index date (maximum up to 15 months); data was retrospectively evaluated over approximately 6 months of this study
Description: Analysis population included all eligible participants whose data were included and observed in this study. AEs were reported as per participants' medical records. There was no specific medical dictionary.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/248
Serious Adverse Events (participants affected / at risk) | 2/248
Other Adverse Events (participants affected / at risk) | 0/248
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=248)
Drug-Drug Interaction (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-03-17): https://cdn.clinicaltrials.gov/large-docs/56/NCT06016556/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-16): https://cdn.clinicaltrials.gov/large-docs/56/NCT06016556/SAP_001.pdf